CLINICAL TRIAL: NCT02268552
Title: An Open Label Multi-part First-in-human Study of Oral LMI070 in Infants With Type 1 Spinal Muscular Atrophy
Brief Title: An Open Label Study of LMI070 (Branaplam) in Type 1 Spinal Muscular Atrophy (SMA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLMI070X2201
Record Dates: First submitted 2014-10-01; First posted 2014-10-20 (Estimated); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: Type 1 Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- branaplam (Experimental): branaplam Treatment
  Interventions: Drug: branaplam

INTERVENTIONS:
Drug: branaplam

SUMMARY:
An open-label, multi-part, first-in-human study of oral branaplam in infants with Type 1 spinal muscular atrophy. The purpose of this study was to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy after 13 weeks; and to estimate the Maximum Tolerated Dose (MTD) of orally administered branaplam; and to identify the dose that was safe for long term use as well as that can provide durable efficacy optimal dosing regimen in patients with Type 1 SMA.

DETAILED DESCRIPTION:
This was an open-label, multi-part, first-in-human, proof of concept study in infants with Type 1 spinal muscular atrophy who have exactly 2 copies of SMN2, to evaluate safety, tolerability, PK, PD and efficacy of oral branaplam after 13 weeks treatment.

Parts 1,2 and 3 were intended to be non-confirmatory.

In Part 1 of the study, patients were dosed once weekly with branaplam. The branaplam dose was escalated in subsequent cohorts until MTD was determined or when sufficient PK results confirmed that the MTD could not be reached due to a potential pharmacokinetic plateau at higher doses. A decision to dose escalate the next cohort was made after safety data was collected for 14 days following the first dose (14-day DLT window). PK was used to confirm that there was no accumulation of the compound. After 13 weeks treatment, participants in part 1 could enter an extension treatment phase until they discontinued from the study or were transferred into part 3.

Part 2 of the study enrolled new patients into one 2 dose cohorts with once weekly dosing for 52 weeks. The branaplam dose was escalated in subsequent cohorts after 6 patients were enrolled and at least 3 patients from the previous cohort completed 13 weeks of treatment. After 52 weeks, patients may have continued treatment in part 3 if it was in the best interest of the patient.

Part 3, participants from part 1 and 2 who have completed at least 52 weeks of banaplam treatment were elegible to continue receiving treatment as long as in the best interest of the patient. In all cases continuation of the treatment was done at a dose selected as optimum, considering existing safety as well as efficacy data.

ELIGIBILITY:
Inclusion Criteria:

Common for both Parts 1 and 2:

* Type 1 SMA, diagnosed clinically, with symptom onset <6 months of age and genetic confirmation of mutations in both alleles of the SMN1 gene, and with SMN2 copy number of 2.
* Best supportive care in place and stable for at least 14 days before screening.
* Must be able to demonstrate antigravity strength in both biceps. At birth gestational age >32 weeks and body weight at birth >2 kg.
* Must live within 2 hours drive of study center. Clearance should be obtained from the site investigator and sponsor if the patient resides more than 2 hours ground travel from the study center

Specific for Part 1

* Age at screening between 1 and 7 months
* Must have or agree to have placement of feeding tube for enteral access via nasogastric (NG), nasojejunal (NJ), percutaneous gastrostomy (PEG), or percutaneous jejunostomy (PEJ) tube for administration of branaplam (for patients in whom branaplam cannot be administered orally ; NG tube may be removed between doses).

Specific for Part 2

* Age at screening between 30 and 180 days of age
* Must have or agree to have placement of feeding tube for enteral access via nasogastric (NG), nasojejunal (NJ), percutaneous gastrostomy (PEG), or percutaneous jejunostomy (PEJ) tube for administration of branaplam (for the first administration only and for patients in whom branaplam cannot be administered orally; NG tube may be removed between doses).
* Minimum CHOP INTEND score of 15 at baseline
* Must be able to feed orally for all nutritional needs and be greater than the 2nd percentile for weight on the standard growth curves for the country of origin

Exclusion Criteria:

Common for both Parts 1 and 2:

* Neurologic, or neuromuscular conditions other than SMA.
* Anemia, leukopenia, neutropenia or thrombocytopenia
* Hepatic dysfunction
* Age adjusted renal dysfunction
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the screening period.
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the screening period.
* Excluding SMA, any medically unstable condition including cardiomyopathy, hepatic dysfunction, kidney disorder, endocrine disorder, GI disorders, prematurity of <32 weeks gestation, metabolic disorders, severe respiratory compromise and significant brain abnormalities or injuries including hypoxic-ischemic encephalopathy.
* Current diagnosis of cardiac and/or vascular abnormalities or ECG abnormalities
* Acute or ongoing medical condition that, according to the Site Investigator and discussed with sponsor, would interfere with the conduct and assessments of the study. Examples are medical disability other than SMA that would interfere with the assessment of safety or would compromise the ability of the subject to undergo study procedures including be assessed by CHOP INTEND motor scale, changes in hematologic parameters or gastrointestinal dysfunction that would compromise the ability of adequate assessment of safety

Specific for Part 1

* Use of other investigational drugs within 14 days.
* Intractable seizure disorder (other than inactive febrile seizures).
* Persistent (in the opinion of the Investigator) hypoxemia (O2 saturation awake <92% or O2 saturation asleep <91%, without ventilation support) or requiring oral suctioning >2 per day, or presence of a tracheostomy.

Specific for Part 2

* Use of nusinersen or gene transfer at any time or other investigational drugs within 14 days.
* Intractable epilepsy
* Persistent (in the opinion of the Investigator) hypoxemia (O2 saturation awake <92% or O2 saturation asleep <91%, without ventilation support), or presence of a tracheostomy.

Ages: 28 Days to 182 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Essen, Germany
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Poland (2):
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Keller CG, Shin Y, Monteys AM, Renaud N, Beibel M, Teider N, Peters T, Faller T, St-Cyr S, Knehr J, Roma G, Reyes A, Hild M, Lukashev D, Theil D, Dales N, Cha JH, Borowsky B, Dolmetsch R, Davidson BL, Sivasankaran R. An orally available, brain penetrant, small molecule lowers huntingtin levels by enhancing pseudoexon inclusion. Nat Commun. 2022 Mar 3;13(1):1150. doi: 10.1038/s41467-022-28653-6. PMID 35241644

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohorts in Part 1 were enrolled sequentially following a 14 day dose-limiting toxicity (DLT) window for each cohort before escalating to the next level. Forty participants were enrolled but only 38 received treatment.
Groups:
- Part 1 LMI070 6mg/m2; Part 1 LMI070 12mg/m2; Part 1 LMI070 24mg/m2; Part 1 LMI070 48mg/m2; Part 1 LMI070 60mg/m2: Single weekly dose for 13 weeks via enteral dosing using nasogastric or nasojejunal or percutaneous endoscopic gastrostomy feeding tubes
- Part 2 LMI070 0.625 mg/kg: LMI070 0.625 mg/kg by enteral route via feeding tube or oral
- Part 2 LMI070 2.5 mg/kg: LMI070 2.5 mg/kg by enteral route via feeding tube or oral
Period: Part 1
Arm/Group | Part 1 LMI070 6mg/m2 | Part 1 LMI070 12mg/m2 | Part 1 LMI070 24mg/m2 | Part 1 LMI070 48mg/m2 | Part 1 LMI070 60mg/m2 | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Started | 2 | 2 | 2 | 4 | 3 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 3 | 0 | 0
Not Completed | 1 | 1 | 1 | 3 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Subject/guardian decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 LMI070 6mg/m2 | Part 1 LMI070 12mg/m2 | Part 1 LMI070 24mg/m2 | Part 1 LMI070 48mg/m2 | Part 1 LMI070 60mg/m2 | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 10 | 15
Completed | 0 (0) | 0 | 0 | 0 | 0 | 10 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 3 Extension
Arm/Group | Part 1 LMI070 6mg/m2 | Part 1 LMI070 12mg/m2 | Part 1 LMI070 24mg/m2 | Part 1 LMI070 48mg/m2 | Part 1 LMI070 60mg/m2 | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Started | 1 | 1 | 1 | 1 | 3 | 10 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1 | 3 | 10 | 12
Not completed — Death | 0 | 1 | 1 | 1 | 1 | 1 | 0
Not completed — Early termination of trial | 1 | 0 | 0 | 0 | 2 | 9 | 11
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1 LMI070 6mg/m2: Enteral dosing using nasogastric or nasojejunal or percutaneous endoscopic gastrostomy feeding tubes for 13 weeks
- Part 1 LMI070 12mg/m2: Single weekly dose for 13 weeks via e teral dosing using nasogastric or nasojejunal or percutaneous endoscopic gastrostomy feeding tubes
- Total: Total of all reporting groups
Arm/Group | Part 1 LMI070 6mg/m2 | Part 1 LMI070 12mg/m2 | Part 1 LMI070 24mg/m2 | Part 1 LMI070 48mg/m2 | Part 1 LMI070 60mg/m2 | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 3 | 10 | 15 | 38
Age, Continuous [Mean (Standard Deviation); unit: months] | 3.0 (1.41) | 4.5 (0.71) | 3.5 (2.12) | 3.8 (1.71) | 5.3 (2.08) | 4.38 (1.521) | 3.81 (1.188) | 4.21 (1.481)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3 | 2 | 5 | 9 | 22
  Male | 1 | 2 | 0 | 1 | 1 | 5 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 2 | 1 | 3 | 2 | 10 | 14 | 34
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Black | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) in Part 1 - Safety Analysis Set (SAS)
Description: A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant therapies that occurs within the first 14 days of treatment with LMI070 and meets any of the criteria for blood and lymphatic system disorders, gastrointestinal disorders, investigations and other toxicities considered clinically significant.
Time Frame: Baseline up to 2 weeks for Part 1
Population: Safety analysis set. No DLTs were observed, therefore maximum tolerated dose could not be determined.
Measure: Number; unit: Participants
Groups:
- Part 1 LMI070 12mg/m2: Enteral dosing using nasogastric or nasojejunal or percutaneous endoscopic gastrostomy feeding tubes for 13 weeks
Arm/Group | Part 1 LMI070 6mg/m2 | Part 1 LMI070 12mg/m2 | Part 1 LMI070 24mg/m2 | Part 1 LMI070 48mg/m2 | Part 1 LMI070 60mg/m2
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events and Deaths- SAS
Description: TEAEs are defined as adverse events starting on or after the first dose of study treatment that were absent pre-treatment, or events present prior to the first dose but increased in severity after the first dose. Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post last treatment.
Time Frame: Baseline up to approximately 83 months
Population: Safety analysis set, all enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 LMI070 6mg/m2 | Part 1 LMI070 12mg/m2 | Part 1 LMI070 24mg/m2 | Part 1 LMI070 48mg/m2 | Part 1 LMI070 60mg/m2 | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 3 | 10 | 15
Participants
  Participants with adverse events | 2 | 2 | 2 | 4 | 3 | 10 | 15
  Participants with serious adverse events | 2 | 2 | 2 | 4 | 3 | 8 | 11
  Deaths | 1 | 2 | 2 | 3 | 1 | 1 | 2

3. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Area Under the Curve (AUCinf) After a Single Dose - Part 1 - Pharmacokinetics Analysis Set (PAS)
Description: The area under the plasma (or serum or blood) concentration-time curve from time zero to infinity [mass x time / volume]
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Part 1 LMI070 Overall: Enteral route via feeding tube or oral. There were 5 cohorts 0.3125, 0.625, 1.25, 2.5, 3.125 mg/kg weekly doses for 2 weeks
Arm/Group | Part 1 LMI070 Overall
Number analyzed (Participants) | 12
h*ng/mL
  0.321 mg/kg - Actual: number analyzed (Participants) | 2
  0.321 mg/kg - Actual | 378 (31.9)
  0.654 mg/kg - Actual: number analyzed (Participants) | 2
  0.654 mg/kg - Actual | 892 (12.3)
  1.39 mg/kg - Actual: number analyzed (Participants) | 1
  1.39 mg/kg - Actual | 1820
  2.49 mg/kg - Actual: number analyzed (Participants) | 4
  2.49 mg/kg - Actual | 3310 (1340)
  2.94 mg/kg - Actual: number analyzed (Participants) | 3
  2.94 mg/kg - Actual | 3800 (1590)

4. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Area Under the Curve (AUCinf) for All Observation Periods - Part 1 - PAS
Description: The area under the plasma (or serum or blood) concentration-time curve from time zero to infinity [mass x time / volume] for all observations. AUC values used for comparison are combined from AUCinf values after single dose and AUC 0-168h values after repeated administration.
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Units Other Than Participants: observations by subject and time point
Arm/Group | Part 1 LMI070 Overall
Number analyzed (Participants) | 13
Number analyzed (observations by subject and time point) | 63
h*ng/mL
  0.299 mg/kg - Actual: number analyzed (observations by subject and time point) | 10
  0.299 mg/kg - Actual | 413 (98.3)
  0.644 mg/kg - Actual: number analyzed (observations by subject and time point) | 4
  0.644 mg/kg - Actual | 761 (170)
  1.30 mg/kg - Actual: number analyzed (observations by subject and time point) | 6
  1.30 mg/kg - Actual | 1340 (381)
  2.52 mg/kg - Actual: number analyzed (observations by subject and time point) | 11
  2.52 mg/kg - Actual | 3310 (850)
  2.95 mg/kg - Actual: number analyzed (observations by subject and time point) | 32
  2.95 mg/kg - Actual | 4210 (1030)

5. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Cmax After a Single Dose - Part 1 - PAS
Description: The observed maximum plasma concentration following drug administration [mass / volume).
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 LMI070 Overall
Number analyzed (Participants) | 12
ng/mL
  0.321 mg/kg - Actual: number analyzed (Participants) | 2
  0.321 mg/kg - Actual | 9.10 (1.22)
  0.654 mg/kg - Actual: number analyzed (Participants) | 2
  0.654 mg/kg - Actual | 18.6 (1.63)
  1.39 mg/kg - Actual: number analyzed (Participants) | 1
  1.39 mg/kg - Actual | 55.6
  2.49 mg/kg - Actual: number analyzed (Participants) | 4
  2.49 mg/kg - Actual | 53.2 (9.50)
  2.94 mg/kg - Actual: number analyzed (Participants) | 3
  2.94 mg/kg - Actual | 72.4 (16.7)

6. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Cmax for All Observation Periods - Part 1 - PAS
Description: The observed maximum plasma (or serum or blood) concentration following drug administration [mass / volume
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: observations by subject and time point
Arm/Group | Part 1 LMI070 Overall
Number analyzed (Participants) | 13
Number analyzed (observations by subject and time point) | 89
ng/mL
  0.299 mg/kg - Actual: number analyzed (observations by subject and time point) | 11
  0.299 mg/kg - Actual | 8.84 (3.58)
  0.644 mg/kg - Actual: number analyzed (observations by subject and time point) | 4
  0.644 mg/kg - Actual | 15.3 (4.10)
  1.30 mg/kg - Actual: number analyzed (observations by subject and time point) | 6
  1.30 mg/kg - Actual | 37.8 (12.8)
  2.51 mg/kg - Actual: number analyzed (observations by subject and time point) | 16
  2.51 mg/kg - Actual | 69.1 (15.7)
  2.95 mg/kg - Actual: number analyzed (observations by subject and time point) | 52
  2.95 mg/kg - Actual | 96.5 (32.7)

7. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Area Under the Curve (AUC) After a Single Dose - Part 2 - PAS
Description: The area under the plasma (or serum or blood) concentration-time curve from time zero to infinity [mass x time / volume)
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Number analyzed (Participants) | 10 | 15
h*ng/mL | 1150 (357) | 4060 (734)

8. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Area Under the Curve (AUC) for All Observation Periods - Part 2 - PAS
Description: The area under the plasma (or serum or blood) concentration-time curve from time zero to infinity [mass x time / volume). AUC values used for comparison are combined from AUCinf values after single dose and AUC0-168h values after repeated administration.
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Units Other Than Participants: observations by subject and time point
Arm/Group | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Number analyzed (Participants) | 10 | 15
Number analyzed (observations by subject and time point) | 28 | 29
h*ng/mL | 1020 (278) | 3470 (909)

9. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Cmax for a Single Dose - Part 2 - PAS
Description: The observed maximum plasma (or serum or blood) concentration following drug administration [mass / volume)
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Number analyzed (Participants) | 10 | 15
ng/mL | 22.0 (5.70) | 82.0 (22.5)

10. Secondary Outcome: Summary of Plasma Pharmacokinetic (PK) Parameter Cmax for All Observation Periods - Part 2 - PAS
Description: The observed maximum plasma (or serum or blood) concentration following drug administration [mass / volume)
Time Frame: from 0 h to 168 h after first/single dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: observations by subject and time point
Arm/Group | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
Number analyzed (Participants) | 10 | 15
Number analyzed (observations by subject and time point) | 29 | 38
ng/mL | 21.7 (5.71) | 77.4 (27.5)

11. Secondary Outcome: Change From Baseline in Growth Parameters: Chest Circumference, Head Circumference and Body Length - Full Analysis Set (FAS)
Description: The effect of branaplam on growth parameters: Length (measured from the top of the head to the sole of the foot), Head circumference and Chest circumference (measured across nipple line). Mean change from baseline in cm is presented
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline, Week 52 and Month 6 of Part 3
Population: Full analysis set - Number of patients who have an assessment available at Baseline and the relevant post-baseline visit.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Parts 1 & 3 Overall; Parts 2 & 3 Overall: Participants who completed 52 weeks of treatment in Part 1 could have continued on same dose or moved to optimal dose (2.5 mg/kg) in Part 3.
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 13 | 25
cm
  Chest - Week 52: number analyzed (Participants) | 10 | 18
  Chest - Week 52 | 4.68 (2.4769) | 5.656 (3.0167)
  Chest - P3 Month 6: number analyzed (Participants) | 6 | 17
  Chest - P3 Month 6 | 14.750 (0548) | 8.582 (2.7423)
  Head -Week 52: number analyzed (Participants) | 10 | 18
  Head -Week 52 | 5.030 (1.1235) | 5.111 (1.3407)
  Head -P3 Month 6: number analyzed (Participants) | 6 | 17
  Head -P3 Month 6 | 9.717 (1.8766) | 6.359 (1.2971)
  Length - Week 52: number analyzed (Participants) | 10 | 19
  Length - Week 52 | 16.950 (3.7825) | 16.942 (4.5806)
  Length - P3 Month 6: number analyzed (Participants) | 5 | 18
  Length - P3 Month 6 | 52.140 (9.8766) | 22.944 (3.7686)

12. Secondary Outcome: Change From Baseline in Growth Parameter: Body Weight - FAS
Description: The effect of Branaplam on body weight in Kg was measured using a weight scale. Mean change from baseline in Kg is presented
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline, Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 13 | 25
kg
  Week 52: number analyzed (Participants) | 10 | 19
  Week 52 | 2.739 (1.3545) | 3.145 (1.5089)
  P3 Month 6: number analyzed (Participants) | 6 | 19
  P3 Month 6 | 9.546 (3.5069) | 4.402 (1.3250)

13. Secondary Outcome: Change From Baseline in Respiratory Function: Pulse Oximetry - FAS
Description: The effect of branaplam on pulse oximetry in percentage of oxygen saturation was evaluated using a probe that measures oxygen in the blood. Mean change from baseline in percentage of oxygen saturation is reported. Negative numbers indicate a decrease from baseline
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline, Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 13 | 25
percentage
  Week 52: number analyzed (Participants) | 9 | 19
  Week 52 | -0.8 (2.59) | -0.1 (1.56)
  P3 Month 6: number analyzed (Participants) | 6 | 19
  P3 Month 6 | -0.7 (2.58) | 0.0 (1.83)

14. Secondary Outcome: Change From Baseline in Respiratory Function: Respiratory Rate - FAS
Description: The effect of branaplam on respiratory rate was evaluated by counting the number of breaths for one minute. Mean change from baseline in breaths per minute is reported"
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline, Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 12 | 25
breaths per minute
  Week 52: number analyzed (Participants) | 8 | 19
  Week 52 | 41.3 (7.57) | 40.5 (13.46)
  P3 Month 6: number analyzed (Participants) | 6 | 18
  P3 Month 6 | 29.2 (6.59) | 37.2 (8.95)

15. Secondary Outcome: Number of Participants With Presence of Paradoxical Breathing - FAS
Description: A paradoxical breathing occurs when one compartment moves out of phase compared to another one.
  In SMA type I, paradoxical breathing is often a sign of breathing problems where the pulmonary ribcage moves inward during inspiration rather than outward while the abdomen expands.
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline, Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 13 | 25
Participants
  Week 52: number analyzed (Participants) | 9 | 19
  Week 52 | 5 | 15
  P3 Month 6: number analyzed (Participants) | 6 | 18
  P3 Month 6 | 4 | 14

16. Secondary Outcome: Change From Baseline in Respiratory Function: Chest Circumference During Quiet Breathing - End of Inspiration and Expiration - FAS
Description: The effect of branaplam on respiratory status was evaluated by measuring the circumference of the ribcage while taking a breathe in and out while quiet or sleeping.
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline, Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 0 | 18
cm
  Week 52 - end of inspiration |  | 5.964 (3.6345)
  P3 Month 6 - end of inspiration: number analyzed (Participants) | 0 | 17
  P3 Month 6 - end of inspiration |  | 8.535 (3.3083)
  Week 52 - end of expiration |  | 6.033 (3.9466)
  P3 Month 6 - end of expiration |  | 9.147 (3.5755)

17. Secondary Outcome: Summary of CHOP INTEND Total Score - Parts 1 and 3 and Parts 2 and 3 - FAS
Description: CHOP INTEND is a motor test measure for SMA Type 1 and similarly weak infants with neuromuscular disease. The CHOP INTEND provides a useful measure of motor skills and strength in this population. It is a 16 item, 64 point scale. Each item (motor skill) is given a score from zero to 4: zero indicates can't complete the movement, 1 to 3 indicates partial performance and a 4 indicates person can complete the movement on their own without assistance. These scores are added up to a possible total score of 64 and higher scores indicate better outcomes.
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline, Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 8 | 18
scores on a scale
  Week 52 | 38.1 (8.69) | 43.6 (6.79)
  Part 3, Month 6: number analyzed (Participants) | 1 | 14
  Part 3, Month 6 | 26.0 | 44.7 (8.73)

18. Secondary Outcome: Number of Participants Fed Orally or by Feeding Tube for Parts 1 and 3 and Parts 2 and 3 - FAS
Description: To evaluate the efficacy of branaplam on preservation of oral feeding
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline up Week 78
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 13 | 25
participants
  Only exclusively orally fed | 3 | 18
  Only exclusively tube fed | 0 | 0
  Started on orally fed, switched to tube fed | 0 | 2
  Started on tube fed, switched to orally fed | 0 | 0
  Other (mixture of both tube and oral feeding) | 8 | 5

19. Secondary Outcome: Number of Participants and HINE Motor Subscale Milestones (Ability to Sit, Stand or Walk Without Support) - FAS
Description: HINE Section 2 is a standardized evaluation of motor function. It evaluates 8 items; grasp, head control, kicking, rolling over, sitting up, crawling, standing and walking. Motor skills are assigned a score of 0 to 3 to 5 points and zero means the child lacks that motor skill. The maximum score is 26 which is dependent on age, level of development and severity of disease. A higher score is a better outcome. This assessment was added with amendment 6, therefore no baseline was available.
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 13 | 25
participants
  Week 52 Sitting - Stable independent sit or Pivots (rotates): number analyzed (Participants) | 3 | 22
  Week 52 Sitting - Stable independent sit or Pivots (rotates) | 1 | 1
  Week 52 Standing - Supports weight: number analyzed (Participants) | 2 | 22
  Week 52 Standing - Supports weight | 0 | 2
  Week 52: Walking - Makes any attempt (i.e., bounces): number analyzed (Participants) | 2 | 16
  Week 52: Walking - Makes any attempt (i.e., bounces) | 0 | 1
  Part 3, Month 6: Sitting - Stable independent sit or Pivots (rotates): number analyzed (Participants) | 5 | 15
  Part 3, Month 6: Sitting - Stable independent sit or Pivots (rotates) | 0 | 4
  Part 3, Month 6: Standing - Supports weight: number analyzed (Participants) | 4 | 15
  Part 3, Month 6: Standing - Supports weight | 0 | 5
  Part 3, Month 6: Walking - Makes any attempt (i.e., bounces): number analyzed (Participants) | 4 | 11
  Part 3, Month 6: Walking - Makes any attempt (i.e., bounces) | 0 | 2

20. Secondary Outcome: Summary of Hammersmith Infant Neurologic Examination Section 2 (HINE-2) - FAS
Description: as for outcome 19
Time Frame: Week 52 and Month 6 of Part 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: total scores
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 5 | 25
total scores
  Week 52: number analyzed (Participants) | 3 | 25
  Week 52 | 3.3 (2.31) | 4.9 (3.44)
  Part 3 Month 6: number analyzed (Participants) | 5 | 15
  Part 3 Month 6 | 3.0 (2.12) | 7.7 (4.82)

21. Secondary Outcome: Ventilation Use for Parts 1 and 3 and Parts 2 and 3 - FAS
Description: BiBAP (bilevel positive airway pressure) ventilation is a 2 level breathing support which has a tube that connects to a mask. It provides a different level of air pressure for inhalation vs. exhalation, whereas a CPAP (continuous positive airway pressure) only pumps one level of air pressure but is also non-invasiive. Invasive ventilation is delivered via an endotracheal or tracheostomy tube.
  In alignment with the study objectives and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration.
Time Frame: Baseline up to 82 months
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Parts 1 & 3 Overall | Parts 2 & 3 Overall
Number analyzed (Participants) | 11 | 25
participants
  Non-invasive ventilation - BiPAP | 9 | 18
  Non-invasive ventilation - CPAP | 3 | 2
  Invasive ventilation | 4 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post last treatment up a maximum of 83 months.
Arm/Group | Part 1 LMI070 6mg/m2 | Part 1 LMI070 12mg/m2 | Part 1 LMI070 24mg/m2 | Part 1 LMI070 48mg/m2 | Part 1 LMI070 60mg/m2 | Part 2 LMI070 0.625 mg/kg | Part 2 LMI070 2.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/2 | 2/2 | 3/4 | 1/3 | 1/10 | 2/15
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 4/4 | 3/3 | 8/10 | 11/15
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 4/4 | 3/3 | 10/10 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 LMI070 6mg/m2 (N=2) | Part 1 LMI070 12mg/m2 (N=2) | Part 1 LMI070 24mg/m2 (N=2) | Part 1 LMI070 48mg/m2 (N=4) | Part 1 LMI070 60mg/m2 (N=3) | Part 2 LMI070 0.625 mg/kg (N=10) | Part 2 LMI070 2.5 mg/kg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 2 | 2 | 4 | 7
Pneumonia aspiration (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0 | 2 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salmonella test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ultrasound kidney abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal tubular disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 LMI070 6mg/m2 (N=2) | Part 1 LMI070 12mg/m2 (N=2) | Part 1 LMI070 24mg/m2 (N=2) | Part 1 LMI070 48mg/m2 (N=4) | Part 1 LMI070 60mg/m2 (N=3) | Part 2 LMI070 0.625 mg/kg (N=10) | Part 2 LMI070 2.5 mg/kg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Reticulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 3
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 3
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heterophoria (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Optic atrophy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2 | 7 | 3
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malocclusion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 3 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Granuloma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical device pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site granuloma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 2 | 2 | 2 | 3 | 7 | 6
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Immunisation reaction (Immune system disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 5 | 8
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 2 | 3
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1 | 1
Ear infection viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 0 | 2 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 0 | 6
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 3 | 3
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 2 | 3 | 2 | 4
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Roseola (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 3 | 4 | 3
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 3 | 2 | 2
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2 | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 5 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Blood iron decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Blood parathyroid hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Body temperature increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 2
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Electrocardiogram P pulmonale (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Heart rate decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Nerve conduction studies abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Reticulocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ultrasound kidney abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 2 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid intake reduced (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Deformity thorax (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rib deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 2 | 4 | 3
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nephrocalcinosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephroptosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 3 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Therapy cessation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tracheostomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cyanosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
In alignment with the study objectives, safety and tolerability of branaplam irrespective of the dose, and protocol defined analyses, secondary efficacy endpoints were analyzed according to the treatment group that participants were assigned at baseline (Part 1&3 and Part 2&3) irrespective of study dose or route of administration. The fact that no dose limiting toxicity was observed in any of the doses and the lack of evidence for dose dependent safety findings further supports this strategy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial

DOCUMENTS (2):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT02268552/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT02268552/SAP_001.pdf